CLINICAL TRIAL: NCT06544083
Title: Early-stage Detection of Liver Cancer by Proteins in Peripheral Blood: a Prospective Study
Brief Title: Early-stage Detection of Liver Cancer by Proteins in Peripheral Blood
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0167
Record Dates: First submitted 2024-04-16; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Diagnosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hepatocellular carcinoma group: Patients with histologically or cytological, imaging confirmed untreated hepatocellular carcinoma.
  Interventions: Diagnostic Test: Proteomics
- Benign liver lesions group: Untreated patients with confirmed or suspected benign liver lesions by histopathology, or with high suspicion of benign liver lesions by imaging evaluation or other routine clinical diagnosis
  Interventions: Diagnostic Test: Proteomics
- Healthy people group: People without any liver disease
  Interventions: Diagnostic Test: Proteomics

INTERVENTIONS:
Diagnostic Test: Proteomics — Proteomic is performed on all blood samples.

SUMMARY:
By collecting blood samples from liver cancer patients and healthy individuals, and comparing the blood protein profiles of the two, the biomarkers for early diagnosis and tissue traceability were identified to accurately establish an early diagnosis model for liver cancer and verify its efficacy.

DETAILED DESCRIPTION:
This study is a prospective study to establish an early diagnosis model for the diagnosis of liver cancer based on peripheral blood protein indexes and verify its efficacy.

The study was divided into two phases: model establishment and model validation. In the model establishment stage, blood samples from subjects with liver cancer and corresponding benign lesions and healthy subjects were prospectively collected, and in the model validation stage, blood samples from subjects with liver cancer and corresponding benign lesions and healthy subjects were included in multiple centers, and a single-blind setting (analyst blinding) was carried out. The diagnosis, follow-up treatment and follow-up of subjects with cancer and benign lesions follow the routine clinical diagnosis and treatment procedures of the research center, and are not affected by this study. Healthy subjects undergo clinical examination in healthy persons according to the protocol of this study. The follow-up diagnosis, treatment and follow-up of subjects judged to be cancer, suspected cancer, benign lesions, and suspected benign lesions during the clinical examination will follow the routine clinical diagnosis and treatment procedures of the research center, and will not be affected by this study. This study is expected to enroll 300 subjects, including 100 subjects with liver cancer, 100 subjects with benign diseases, and 100 healthy subjects. The study is divided into two phases, and the first phase of the study will enroll 150 subjects, including 50 subjects with liver cancer, 50 subjects with benign disease, and 50 healthy subjects. The second phase of the study will enroll 150 subjects, including 50 cancer subjects, 50 benign disease subjects, and 50 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent.
2. Male or female, age equal to or greater than 18 years and less than 75 years.
3. Patients with liver cancer who have been diagnosed or suspected for the first time within 42 days prior to blood collection
4. The subject has not undergone any local or systemic anti-tumor therapy before blood collection, including (but not limited to) tumor surgical treatment for any purpose, local or systemic chemoradiotherapy, targeted therapy (including anti-angiogenic drugs), immunotherapy, cancer vaccine and hormone therapy, etc.
5. Patients with histologically or cytological, radiographically confirmed hepatocellular carcinoma.

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding.
2. Previous organ transplantation or non-autologous bone marrow or stem cell transplantation.
3. Received drugs with anti-tumor effects for other diseases within 30 days before blood collection, such as drugs used for the treatment of immunorheumatic diseases such as methotrexate, cyclophosphamide, thiazoprine, chlorambucil, etc., drugs for the treatment of breast diseases, such as tamoxifen, etc.
4. History of previous malignant tumors.
5. Having other malignant tumors or multiple primary tumors at the same time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female, aged 18 years or older, less than 75 years of age and people who voluntarily sign informed consent
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood protein concentrations | up to 2 years
  The blood of liver cancer patients before treatment and the blood of non-liver cancer subjects were collected, and the differences between the peripheral blood protein characteristics of the above groups and those of non-liver cancer subjects and the blood protein characteristics that can be used for tissue traceability were analyzed. Peripheral blood protein concentrations were quantitatively measured by proteomic methods. Univariate COX regression method will be used to analyze whether the differences between the two groups are related to the diagnosis of liver cancer.
An early diagnosis model of liver cancer | up to 2 years
  The sensitivity and specificity of an early diagnosis model for the diagnosis of liver cancer based on peripheral blood protein indexes and the accuracy of tissue traceability were established and verified.

SECONDARY OUTCOMES:
Presence or absence of intrahepatic and extrahepatic metastases of liver cancer | up to 2 years
  The number and size of intrahepatic and extrahepatic metastases of liver cancer were measured by imaging methods to evaluate whether they were associated with the high risk predicted by the diagnostic model of liver cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Weilin Wang, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Yuan Ding, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Zhongquan Sun, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided